CLINICAL TRIAL: NCT02569762
Title: Assessment of the Effect of Artificial Sweeteners on Gut Microbiota and Glucose Metabolism
Brief Title: Effects of Artificial Sweeteners on Gut Microbiota and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2015:069
Record Dates: First submitted 2015-07-21; First posted 2015-10-07 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-05

CONDITIONS: Impaired Glucose Tolerance
Keywords: Non-Nutritive Sweeteners; Artificial Sweeteners; Glucose Metabolism; Microbiota; Dysbiosis
MeSH Terms: conditions — Glucose Intolerance; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucralose-Aspartame (Experimental): Generic name: sucralose or aspartame, Dosage form: powder, Duration:seven days.
  Interventions: Dietary Supplement: Sucralose-Aspartame; Dietary Supplement: Aspartame-Sucralose
- Aspartame-Sucralose (Experimental): Generic name: aspartame or sucralose, Dosage form: powder, Duration:seven days.
  Interventions: Dietary Supplement: Sucralose-Aspartame; Dietary Supplement: Aspartame-Sucralose

INTERVENTIONS:
Dietary Supplement: Sucralose-Aspartame — Sucralose or aspartame
Dietary Supplement: Aspartame-Sucralose — Aspartame or sucralose

SUMMARY:
The Objectives of this study is to determine the effect(s) of daily non-caloric artificial sweetener (NAS) consumption (sucralose or aspartame) on the composition of the bacteria and also to determine the changes in glucose metabolism.

DETAILED DESCRIPTION:
The trial will be 12 weeks randomized, cross-over and double blinded with 2 treatment intervention ( sucralose and aspartame) , there will be a run in period (4 weeks), then phase 1 treatment period for two weeks followed by four weeks washout period then phase 2 treatment period(2 weeks). Healthy, normglycemic (<5.6 mmol/L) males and females ( 17 total) of age 18-45 y with a body mass index (BMI) 20-25 kg/m2 will be recruited.

Each participants will be given the dose of sweetener aspartame or sucralose during the treatment phase in a double-blind procedure.

the participant will be asked to consume the sweetener in a mixed flavoured beverage during each visit in the treatment phase.

Blood and stool sample collection will take place before after the run-in period, and after the washout period, as well as after each two-week treatment period.

glucose measurement: Capillary blood will be collected during each visit by registered nurse. Blood will be collected at fasting and at 12,30,45,60,90 and 120 minutes after the participants drink a glucose drink (75g glucose) for Oral glucose tolerance test.

a food frequency questionnaire will be given to each participant in order to estimate how often each sweetener is consumed on a daily basis.

Participants will also be asked to complete weekly food diaries of food and drink consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20-25 kg/m2
* Fasting blood glucose (FBG) < 5.7 mmol/L
* women with regular menstrual cycle.

Exclusion Criteria:

* probiotic or antibiotic use within 6 months prior to the start of the study
* metabolic or gastrointestinal disorders (diabetes mellitus types 1 and 2, inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), celiac disease, phenylketonuria)
* pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | 0-200 mins
  Fasting blood glucose level and 2-hour oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Insulin, glucagon,GIP & GLP-1 | 4 times during the 12 weeks period
  glucose homeostasis
Fecal Microbiome & short chain fatty acids measurements | 4 times during the 12 weeks period
  to detect bacterial composition in feces and SCFA changes

CONTACTS AND LOCATIONS:
Overall Officials: James K Friel, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods & Nutraceuticals, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided